CLINICAL TRIAL: NCT00081913
Title: Injection of Autologous CD34-Positive Cells for Neovascularization and Symptom Relief in Patients With Myocardial Ischemia
Brief Title: Stem Cell Study for Patients With Heart Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Losordo, Douglas, M.D. (Individual)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 00165
Record Dates: First submitted 2004-04-26; First posted 2004-04-28 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Chest Pain; Myocardial Ischemia; Heart Disease; Coronary Arterial Disease (CAD); Angina
Keywords: Apheresis; Cell Transfer; Chest Pain; Adult Stem Cell Therapy
MeSH Terms: conditions — Chest Pain; Myocardial Ischemia; Heart Diseases; Angina Pectoris

INTERVENTIONS:
Genetic: Cell Therapy - Autologous CD34 Positive Cells

SUMMARY:
The purpose of this study is to determine if cell therapy with your own cells (autologous cells) delivered with a catheter to regions of the heart with poor blood flow will be safe and if it will relieve your chest pain and/or your ability to exercise.

DETAILED DESCRIPTION:
The goal of this study is to determine the safety of various doses of autologous (one's own) stem cells, delivered with a catheter into the regions of the heart with poor blood flow. Stem cells are primitive cells produced by bone marrow that can develop into blood cells or other types of cells. In addition to determining whether this new approach is safe, the diagnostic tests may offer preliminary insights into the usefulness of this approach for treating myocardial ischemia (the condition where areas in the heart are lacking enough oxygen and blood flow to keep the heart muscle working well).

This is a blinded, randomized study to compare a certain type of stem cell called CD34-positive versus a placebo agent (normal saline). You will have a 3:1 chance of receiving your CD34-positive stem cells versus the placebo agent (normal saline). You will not know whether you received the CD34-positive cells or the placebo agent (normal saline). If you are randomized to receive placebo (normal saline), you will undergo all of the pre-treatment phases of this study (including the stem cell mobilization phase and the apheresis procedure), but rather than receiving injections of CD34-positive cells, you will receive injections of the placebo agent (normal saline). There is some research evidence that suggests CD34-positive cells may help develop new blood vessels or improve blood flow when injected directly into the heart muscle.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with functional class (CCS) III or IV angina.
* Subjects who have attempted "best" medical therapy without control of symptoms.
* All subjects must have a recent coronary angiogram (within the last 3 months).
* Clinical signs and symptoms of clinically significant ischemia on nuclear perfusion imaging.
* Subjects must be able to complete a minimum of 1 minute but no more than 6 minutes of the Standard Bruce Protocol.
* Subject experiences angina during the baseline exercise tolerance test.
* Subjects must either be no longer capable of reproduction or taking acceptable measures to prevent reproduction during the study.
* Normal renal function.
* Normal liver function.
* Normal blood count.

Angiographic Inclusions:

* Total occlusion of an epicardial coronary artery.
* Candidates at high risk for percutaneous coronary angioplasty of treatment zone(s) based upon clinical or anatomic considerations including but not limited to the following: diabetes, congestive heart failure (severe right heart failure, NYHA class III or IV), left main disease, pulmonary hypertension, severe proximal vessel tortuosity, severe bendpoint obstructions, diffuse disease (>2 cm in length), small vessel (<2 mm reference diameter), stenosis which are either diffuse (>2 cm in length) or distal, incessant restenosis lesions, unfavorable bifurcation stenosis, and degenerated or thrombosed saphenous vein grafts.

Exclusion Criteria:

* Predominant congestive heart failure symptoms.
* Patients who have been hospitalized with a primary diagnosis of CHF in the prior 6 months.
* Patients who have had diuretics added to their medical regimen or an increase in diuretic dosage for signs or symptoms of CHF in the past 6 months.
* Patients with a left ventricular ejection fraction of less than 25% as determined by transthoracic echocardiography.
* Patients with physical findings consistent with ongoing uncontrolled CHF.
* Myocardial infarction within 30 days of treatment.
* Successful coronary revascularization procedures within 3 months of study enrollment.
* Documented stroke or transient ischemic attack (TIA) within 60 days of study enrollment.
* History of severe aortic stenosis or insufficiency; severe mitral stenosis; or severe mitral insufficiency.
* Severe co-morbidity associated with a reduction in life expectancy of less than 1 year.
* Subjects with PT, PTT or platelet counts greater than the upper limit of normal and those with a hematocrit <35%.
* Subjects with uncontrolled hypertension.
* Currently enrolled in another investigational device or drug trial (IDE or IND) that has not completed the required follow-up period.
* History of alcohol or drug abuse within 3 months of screening.
* Joint or peripheral vascular disease that severely limits treadmill walking.
* Chronic obstructive pulmonary disease that severely limits walking or FEV1.0<30% predicted.
* Subjects who are pregnant or lactating.
* Males and females who are capable of reproduction and will not take acceptable measures to prevent reproduction during the study.
* Subjects who test positive for HIV, hepatitis B or hepatitis C, have a chronic inflammatory disease, autoimmune disease or are on chronic immunosuppressive medications.
* Subjects with a known hypersensitivity to E. coli-derived proteins.
* Subjects with evidence (clinical, laboratory, or imaging) of cancer recurrence within the past 5 years (other than non-melanoma skin cancer or in situ cervical carcinoma).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2004-01; Primary Completion 2006-03 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Scripps Clinic, La Jolla, California
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota

REFERENCES:
- [Derived] Losordo DW, Schatz RA, White CJ, Udelson JE, Veereshwarayya V, Durgin M, Poh KK, Weinstein R, Kearney M, Chaudhry M, Burg A, Eaton L, Heyd L, Thorne T, Shturman L, Hoffmeister P, Story K, Zak V, Dowling D, Traverse JH, Olson RE, Flanagan J, Sodano D, Murayama T, Kawamoto A, Kusano KF, Wollins J, Welt F, Shah P, Soukas P, Asahara T, Henry TD. Intramyocardial transplantation of autologous CD34+ stem cells for intractable angina: a phase I/IIa double-blind, randomized controlled trial. Circulation. 2007 Jun 26;115(25):3165-72. doi: 10.1161/CIRCULATIONAHA.106.687376. Epub 2007 Jun 11. PMID 17562958
- See also: Caritas St. Elizabeth's Medical Center of Boston — http://www.semc.org